CLINICAL TRIAL: NCT02156817
Title: Neurophysiologic Maturation Index: NEMO Project for Late Preterm Infants
Brief Title: Neurophysiologic Maturation Index for Late Preterm Infants
Acronym: NEMO Project
Status: Completed | Type: Observational
Sponsor: Brown University (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Birju A. Shah, MD MPH, Associate Professor of Pediatrics, University of Oklahoma
Other Study IDs: 13-0052
Record Dates: First submitted 2014-05-17; First posted 2014-06-05 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Neurophysiologic Maturation
Keywords: Amplitude integrated electroencephalogram; Heart rate variability; Respiratory rate variability; Preterm Infants; Length of Hospital Stay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Late Preterm Infants (LPT): 34 weeks and 0-6 days gestational age
  Interventions: Other: Amplitude integrated electroencephalogram, Cardiorespiratory signal acquisition

INTERVENTIONS:
Other: Amplitude integrated electroencephalogram, Cardiorespiratory signal acquisition

SUMMARY:
Late preterm infants contribute to significant neonatal intensive care unit health care resource utilization because of their sheer numbers. Determinants of the length of hospitalization (LOH) in this population are understudied. Gestational age (GA) is used most commonly as a predictor for LOH but there are many limitations including inaccurate dating and morbidities of prematurity which at least partly related to neurophysiological immaturity. The latter can be assessed by amplitude integrated electroencephalogram (aEEG, a simplified 5 lead EEG), and possibly by heart rate variability (HRV) and respiratory variability (RV). All 3 are non-invasive tests that can be done at the bedside. Our study hypothesis is to determine if neurophysiologic maturation as assessed by aEEG, HRV and RV within 24-96 hours following birth improves the correlation between gestational age and length of hospitalization compared to gestational age alone.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 340-346 weeks by Obstetric criteria (presence of a sure LMP or sonogram performed in the first trimester, or agreement between LMP and a sonogram performed between the first trimester and 20 weeks)
* Admitted to a NICU of a participating institution
* Post-natal age less than 96 hours

Exclusion Criteria:

* Major congenital anomaly/genetic anomaly
* Growth restriction (birth weight < 10%, Fenton growth curves)
* Unsure obstetric dating (e.g., absence of a sure LMP without a sonogram, earliest sonogram performed after 20 weeks without a sure LMP, or discrepancy between LMP and sonogram)
* Exposure to medications within the preceding 12 hrs which may affect CNS function (e.g., fentanyl, morphine, midazolam)
* Neonatal seizures
* Neonatal abstinence syndrome secondary to in-utero exposure to narcotics, methadone etc, or at high risk for development of abstinence
* Hypoxia-ischemia defined as the combination of fetal acidemia (cord gas or blood gas within 1 hour of birth: pH ≤ 7.15 or BE ≥ -10mEq/L), need for resuscitation at birth (PPV ± chest compressions or medications), and evidence of encephalopathy (Stage 1, 2 or 3 Sarnat). Stage 1 encephalopathy will be defined based on the level of consciousness which is characterized by a hyper-alert state, apparent alertness, and irritability. In the absence of a cord or early post-natal blood gas, there must be a history of a perinatal event which may have compromised oxygenation or blood flow to the fetus.
* Infants who are expected to be on mechanical (via an endotracheal tube) or high frequency ventilation for the first 96 hours after birth.
* Inability to obtain the informed consent

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal intensive care unit Newborn nursery
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08-18 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Magnitude of variance, R square | 2 years
  linear regression model: LOH = intercept + b1GA + b2aEEG + b3HRV + b4RV + error term; b1 - b4 represents the weight of each variable to explain the variance of the equation (R2), GA is gestational age, aEEG is amplitude integrated EEG, HRV is heart rate variability, RV is respiratory variability, LOH is length of hospital stay

SECONDARY OUTCOMES:
Amplitude integrated electroencephalogram (aEEG) | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  number of cycles/hour, the lower border voltage, the span voltage or the percent of the tracing which is discontinuous
Heart rate variability (HRV) | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  standard deviation of the R-R interval, sample asymmetry and sample entropy
Respiratory variability (RV) | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  instantaneous respiratory effort, phase between ribcage and abdomen, amplitude of the signal, pause metrics and movement artifact metrics

CONTACTS AND LOCATIONS:
Overall Officials: Birju A Shah, MD, MPH, Principal Investigator — Brown University - Women and Infants Hospital of Rhode Island; Abbot Laptook, MD, Principal Investigator — Brown University - Women and Infants Hospital of Rhode Island
Locations (3):
- United States (2):
  - Wayne State University, Detroit, Michigan
  - Brown University - Women and Infants Hospital of Rhode Island NICU, Providence, Rhode Island
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Background] Shah BA, Latremouille S, Chawla S, Keszler M, Tucker R, Laptook A, Sant'anna GM. Heart rate variability and amplitude-integrated electroencephalography measured shortly after birth and time to reach clinical milestones: a pilot study in late preterm infants. Front Pediatr. 2025 Jun 5;13:1579197. doi: 10.3389/fped.2025.1579197. eCollection 2025. PMID 40538931